CLINICAL TRIAL: NCT02101645
Title: Proof-of-concept Study for Bioimpedance Based Monitoring of Venous Ulcers During Galvanic Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other); Åbo Akademi University (Other); Aalto University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: R13148
Record Dates: First submitted 2014-02-26; First posted 2014-04-02 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Patients With Lower Extremity Venous Ulcers; Patients With Localized Edema
Keywords: Bioimpedance; Venous ulcer; Edema; LIDC; Electrical stimulation
MeSH Terms: conditions — Varicose Ulcer; Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LIDC treatment and bioimpedance monitoring of venous ulcers. (Experimental): Lower extremity venous ulcers will be treated using periodical LIDC stimulation. Wound healing and edema reduction efforts will be monitored using bioimpedance based monitoring.
  Interventions: Procedure: Periodical low intensity direct current (LIDC) stimulation of wound.; Procedure: Compression therapy of swollen limbs.

INTERVENTIONS:
Procedure: Periodical low intensity direct current (LIDC) stimulation of wound. — Wound is stimulated using LIDC current. Stimulation current magnitude is in micro-ampere range. Stimulation sequence is 1 hour on and 1 hour off for 72 hours or 96 hours.
Procedure: Compression therapy of swollen limbs. — Compression bandage is used for reducing swelling of the limbs.

SUMMARY:
The research group will choose no more than 10 patients having a lower extremity venous ulcer(s), less than 5cm diameter and with an estimated one month time of re-epithelization. In this study the investigators will follow and monitor the healing of the wound and effectiveness of compression therapy using bioimpedance measurement based method. The investigators will also treat the wounds using periodical low intensity direct current (LIDC) stimulation therapy.

Bioimpedance monitoring and wound stimulation functionalities are provided by a purpose built wound patch. The patch features a printed 4 x 4 stimulation and impedance measurement electrodes array (in contact with wound surface) surrounded by a 4-part dual purpose counter and impedance reference electrodes (in contact with the intact skin surrounding the wound area).

DETAILED DESCRIPTION:
Objectives of the study

Primary: Proof-of-concept study of bioimpedance measurement based method for monitoring of chronic wound healing and assessment of efficacy of compression therapy. Gathering bioimpedance data from the patients with a lower extremity ulcer of venous etiology over their healing process. The investigators will seek methods for processing the collected data to find the best correlation with visually observed healing of the wound.

Secondary: Proof-of-concept study of periodical LIDC wound stimulation. The investigators will compare the LIDC enhanced healing outcome with appropriate archived data of previous studies performed in TAYS.

Other: Analysis of the received data and reliability evaluation of the methods. Gathering relevant user feedback from medical personnel and patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with a chronic wound of venous origin.
* Patients have signed consent to participate in the study.
* Patient is motivated to follow the instructions given by medical personnel and research group.
* Age 18 - 80 years.
* Wound(s) is expected to heal significantly during the period of 2 months.
* Wound(s) is located so that there is enough space to place the experimental wound dressing appropriately.
* Diameter of a single wound is no more than 5 cm and wound edges are not steep. If patient has multiple small wounds, the wounds are located within an area of 5x5cm.
* Patient has adequate vascular supply and patient tolerates compression dressings.

Exclusion Criteria:

* Patient has an unstable coronary disease.
* Subject does not approve the informed consent.
* Subject is not appropriately motivated to follow M.D.'s instructions of treatment (at home).
* Participation in another clinical trial that involves an investigational drug or device that would interfere this study.
* Patient suffers from cognitive problem such as dementia.
* Wound is not expected to be healed during the time reserved for the measurements (circa 2 months).
* Patient has active wound infection or increased risk of wound infection.
* Skin changes or skin disease which could alter the epidermis of the electrode site during the measurement period.
* Patient has cancer or other life threatening disease in an unstable condition.
* Patient is pregnant.
* Patients with implantable electrical device. Such as pacemaker or implanted defibrillator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
2-electrode bioimpedance data of wound and intact skin. 4-electrode bioimpedance data related to local interstitial fluid status of affected leg. | 4 months
  We aim to determine how well bioimpedance measurement based method for monitoring of chronic wound healing and assessment of efficacy of compression therapy comply with the results of conventional wound monitoring methods.
  We will measure the impedance of the wound and intact skin from multiple locations using 2-electrode configuration. To obtain this a purpose built electrode array will be placed on the wound, covering also area of intact skin. The electrode array will also be used for determining the interstitial fluid status of the leg by 4-electrode impedance measurement.

SECONDARY OUTCOMES:
Low intensity direct current stimulation of wound. | 4 months
  We will compare the LIDC enhanced healing outcome with appropriate archived data of previous studies performed in Tampere University Hospital.

OTHER OUTCOMES:
Patient and personnel questionaire results. | 2 months
  After the final patient visit, a questionaire will be given to patients and personnel. Questionaire will provide the research group valuable information for further development of the study method and equipment.

CONTACTS AND LOCATIONS:
Overall Officials: Annikki Vaalasti, MD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

REFERENCES:
- [Result] Ward L, Winall A, Isenring E, Hills A, Czerniec S, Dylke E, Kilbreath S. Assessment of bilateral limb lymphedema by bioelectrical impedance spectroscopy. Int J Gynecol Cancer. 2011 Feb;21(2):409-18. doi: 10.1097/IGC.0b013e31820866e1. PMID 21270623
- [Result] Carley PJ, Wainapel SF. Electrotherapy for acceleration of wound healing: low intensity direct current. Arch Phys Med Rehabil. 1985 Jul;66(7):443-6. PMID 3893385
- [Result] Zhao M, Song B, Pu J, Wada T, Reid B, Tai G, Wang F, Guo A, Walczysko P, Gu Y, Sasaki T, Suzuki A, Forrester JV, Bourne HR, Devreotes PN, McCaig CD, Penninger JM. Electrical signals control wound healing through phosphatidylinositol-3-OH kinase-gamma and PTEN. Nature. 2006 Jul 27;442(7101):457-60. doi: 10.1038/nature04925. PMID 16871217
- [Result] Blount AL, Foster S, Rapp DA, Wilcox R. The use of bioelectric dressings in skin graft harvest sites: a prospective case series. J Burn Care Res. 2012 May-Jun;33(3):354-7. doi: 10.1097/BCR.0b013e31823356e4. PMID 21979844
- [Result] Weber SA, Gehin C, Moddy G, Jossinet J, McAdams ET. Characterisation of a multi-frequency wound impedance mapping instrument. Annu Int Conf IEEE Eng Med Biol Soc. 2008;2008:4907-10. doi: 10.1109/IEMBS.2008.4650314. PMID 19163817
- See also: Micro-current treatment dressing for chronic wounds — http://procellera.com/